CLINICAL TRIAL: NCT04552171
Title: Game Plan: Testing the Efficacy of a Brief, Web-based Intervention in Reducing Heavy Drinking and Reducing Sexually-transmitted Infections Among High-risk Men Completing Self-testing
Brief Title: Game Plan: Efficacy of a Brief, Web-based Intervention on Alcohol Use and Sexually-transmitted Infections
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2003002671
Record Dates: First submitted 2020-08-28; First posted 2020-09-17 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Sexually Transmitted Diseases, Bacterial; Alcohol; Harmful Use
MeSH Terms: conditions — Sexually Transmitted Diseases, Bacterial

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned 1:1 to one of two conditions: (1) a 24-hour helpline providing free standard post-test counseling and referral, or (2) the 24-hour helpline plus the Game Plan app. In both conditions, participants will be encouraged to use these services via a large postcard included in each test kit and via email, and so, can use them after each test.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All key study personnel will be blinded to participants' condition assignments. Since participants are encouraged to complete both STI self-testing and follow-up online surveys via automated emails linking to a web-based survey system, no members of the study staff will be serving as outcomes assessors. As such, outcomes assessment is also blinded to study condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to Game Plan app and 24-hour helpline (Experimental): Participants in this condition will be provided access to the Game Plan app and encouraged to use it after they complete their baseline assessments and STI testing has been completed. These participants will also be provided with access to a 24-hour helpline that provides free HIV/STI test counseling, which they can elect to use or not.
  Interventions: Behavioral: Access to Game Plan app and 24-hour helpline
- Access to a 24-hour helpline (No Intervention): Participants in this condition will be provided access to a 24-hour helpline that provides free HIV/STI test counseling, which they can elect to use or not. Use of this comparison condition is intended to provide a real-world test of the added benefit of using Game Plan, above and beyond the current "standard of care" for HIV/STI self-testing, which involves providing users with access to a 24-hour helpline.

INTERVENTIONS:
Behavioral: Access to Game Plan app and 24-hour helpline — Game Plan is a web-based application that helps users reflect on their risk for HIV and level of alcohol use, and if interested, make a plan for reducing their sexual risk or drinking.
  Arms: Access to Game Plan app and 24-hour helpline

SUMMARY:
The proposed study involves conducting a larger-scale study exploring Game Plan's effects among MSM in the real-world, alongside innovative approaches for expanding HIV testing. Using a hybrid 1 effectiveness-implementation approach, the investigators will recruit up to 360 high-risk, heavy drinking MSM online from several high-incidence areas in the US to participate in a program providing home-based HIV/STI self-tests in the mail at regular intervals over a year (baseline, 6 months, 12 months). Participants will be randomly assigned to receive access to either (1) a 24-hour helpline for counseling/referrals, or (2) the helpline plus Game Plan. Investigators will test whether those who use Game Plan show lower rates of heavy drinking, any STIs, and high-risk CAS events compared to those receiving access to the helpline alone.

DETAILED DESCRIPTION:
This is a hybrid 1 effectiveness-implementation, mixed methods study that involves conducting a longitudinal randomized controlled trial in which high-risk, heavy drinking MSM (N = 360) will be recruited online from several high-incidence US cities: Atlanta, Los Angeles, Miami, New Orleans, Washington DC/Baltimore. Participants will be sent HIV and STI self-testing kits at baseline, 6 mo., and 12 mo. Along with their test kits, they will be randomized to receive access to either: (1) a 24-hour helpline providing free standard post-test counseling and referral, or (2) the 24-hour helpline plus the Game Plan app. Test kits will provide testing and results for HIV, Syphilis, and genital, rectal, and pharyngeal Gonorrhea and Chlamydia, as well as phosphatidylethanol (PEth). Participants will also be asked to complete an online follow-up survey every three months that assess drinking, sexual behavior, and use of prevention methods over the 12-month study period. At 12 mo., 30 participants and 12 HST stakeholders will be recruited to participate in qualitative interviews to issues relevant to implementing Game Plan alongside HIV testing programs. Specifically, this study aims to: (1) test whether using a brief, MI-inspired, web-based intervention (Game Plan) after HST reduces (a) binge drinking, (b) the average number of drinks per drinking day over 12 months among heavy-drinking and high-risk, HIV-negative MSM, compared to providing access to a 24h helpline providing risk-reduction counseling alone, (2) test whether using Game Plan results in lower rates of (a) bacterial STIs, (b) high-risk CAS, and (c) higher rates of PrEP uptake over 12 months, and (3) to assess Game Plan's potential for implementation into self-testing programs by examining indicators of adoption, engagement, appropriateness and satisfaction among MSM assigned to have access to the site. Investigators will use site metrics and responses, survey data, and in-depth qualitative interview data from users and virtual focus groups with stakeholders to help address key implementation questions.

ELIGIBILITY:
Inclusion Criteria:

* Assigned male sex at birth
* Currently male gender
* 18+ years old
* HIV-negative or unknown status
* Able to speak and read English or Spanish fluently
* Report drinking heavily within the past month, defined according to NIAAA guidelines as having drank >5 drinks on a single occasion at least once or an average of >14 drinks in a given week
* Not being currently prescribed or taking PrEP
* Having met at least one of three HIV-risk-related PrEP eligibility criteria in the last 6 months: (a) having been diagnosed with an STI, (b) currently having regular anal sex with a man who is HIV-positive, or (c) having had anal sex without a condom with a man outside of the context of a sexually exclusive relationship with a single partner who has been recently tested and is HIV-negative.

Exclusion Criteria:

* Injection drug use in the past year
* Screened positive for drug use disorder
* Report history or risk of complicated alcohol withdrawal
* Report currently receiving medications or counseling for an alcohol or drug use disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants who are (1) assigned male sex at birth, and (2) currently male gender are eligible.
Enrollment: 500 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of alcohol drinking days in the past 30 days | 3 months, 6 months, 9 months, 12 months
  Total number of days in which participants reported drinking over the 30 days preceding each follow-up
Number of heavy (5+ standard drinks) alcohol drinking days in the past 30 days | 3 months, 6 months, 9 months, 12 months
  Total number of days on which participants reported consuming 5+ standard drinks in a given day over the 30 days preceding each follow-up
Average number of standard drinks consumed on a drinking day in the past 30 days | 3 months, 6 months, 9 months, 12 months
  The average number of standard drinks participants reported consuming when they drank over the 30 days preceding each follow-up
Any new bacterial sexually-transmitted infection diagnosis | 6 months, 12 months
  Whether or not participants were diagnosed with a bacterial sexually-transmitted infection (Chlamydia or Gonorrhea at genital, oral, or rectal sites, or Syphilis) in the past 6 months
Number of sex events that pose risk for sexually-transmitted infections in the past 30 days | 3 months, 6 months, 9 months, 12 months
  The total number of sex events in which participants reported engaging in insertive or receptive anal sex with a non-exclusive partner or partner whose HIV status is uncertain without using a condom, or for those who have started PrEP, without reporting having taken a dose within 2 days of sex occurring, in the 30 days preceding each follow-up
Receiving a prescription for pre-exposure prophylaxis | 6 months, 12 months
  Whether or not participants reported receiving a prescription for pre-exposure prophylaxis in the 6 months prior to each follow-up

SECONDARY OUTCOMES:
HIV diagnosis | 6 months, 12 months
  Whether or not participants were diagnosed with HIV at any time during the 12-month study period
Phosphatidylethanol quantity | 6 months, 12 months
  The quantity of phosphatidylethanol detected in dried blood spots collected at 6- and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Tyler B Wray, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be uploaded to the National Institute on Alcohol Abuse and Alcoholism data archive (NIAAA-DA) every 6 months while the trial is actively recruiting and collecting data, with a final dataset planned for upload within 6 months of the final follow-ups being conducted, as per NIAAA policy. The dataset will be formatted, structured, and curated to align with NIAAA policy.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Full datasets of participants agreeing to share their data with the NIAAA-DA will be uploaded once every 6 months while the trial is ongoing, with a final dataset uploaded within 6 months of completing the final follow-ups. Data will be made available from the NIAAA-DA for registered researchers after an embargo period of 2 years after the final dataset is uploaded.
Access Criteria: Researchers who have registered with the NIAAA-DA are eligible to access data from this trial.
URL: https://www.niaaa.nih.gov/research/niaaa-data-archive

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT04552171/Prot_SAP_000.pdf